CLINICAL TRIAL: NCT02253810
Title: The Effect of Intravenous Tranexamic Acid on Blood Loss and Transfusion After Periacetabular Osteotomy: a Prospective, Double-blinded, Randomized Controlled Trial
Brief Title: Efficacy of Tranexamic Acid for Reducing Blood Loss and Blood Transfusion After Periacetabular Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-115
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Dysplasia, Congenital Hip
Keywords: Dysplasia, Congenital Hip; Osteotomy; Blood Transfusion; Tranexamic Acid
MeSH Terms: conditions — Hip Dislocation, Congenital | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Patients randomized to this arm will receive standard dosing of tranexamic acid intraoperatively.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Patients randomized to this arm will receive normal saline solution, instead of tranexamic acid, intraoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Medication administered intra-operatively to promote blood clotting.
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Placebo — Saline solution
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled, double-blinded trial is to assess the efficacy of intravenous tranexamic acid, a drug, in reducing blood loss and transfusion in patients undergoing periacetabular osteotomy, an elective reorientation procedure for the hip joint. The investigators hypothesize that tranexamic acid will be more effective than placebo (normal saline solution) in reducing blood loss and transfusion after periacetabular osteotomy.

DETAILED DESCRIPTION:
Periacetabular osteotomy (PAO) is an elective reorientation surgery for the hip joint, typically for the treatment of hip dysplasia in young, otherwise healthy patients, which requires multiple pelvic osteotomies around the acetabulum. A major source of its perioperative morbidity is blood loss. The principal cause of postoperative blood loss after PAO is surgical trauma, with secondary activation of both the coagulation cascade and local fibrinolysis. In the PAO literature, allogeneic transfusion rates are as high as 58%, and blood loss can range to nearly 4 L. The risk of excessive blood loss and blood transfusion in young, healthy patients after elective surgery is an event that can be reduced with blood conservation protocols, which can include pharmacological agents. Tranexamic acid is a synthetic derivative of the amino acid lysine and a competitive inhibitor of plasminogen activation that interferes with fibrinolysis. Multiple studies and meta-analyses have shown that intravenous administration of the antifibrinolytic agent tranexamic acid reduces postoperative bleeding and the need for transfusion during joint replacement surgery. However, no published data exists to support its use during PAO. We hypothesize that intravenous tranexamic acid will reduce perioperative blood loss and, thus, transfusion requirement in patients undergoing PAO. A total of 80 patients will be enrolled. Patients will be randomized to receive either intravenous tranexamic acid versus placebo (normal saline) during PAO. Calculated total blood loss (primary outcome) will be determined, and intraoperative cell saver utilization (secondary outcome), and (3) postoperative allogeneic blood transfusion (secondary outcome) will be recorded. Patients will be followed for a total of 6 weeks after surgical intervention. If the use of IV tranexamic acid in the PAO patient population significantly reduces total perioperative blood loss, then it would provide an efficacious and inexpensive method for reducing postoperative morbidity after PAO.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 12 years old
* Age less than or equal to 45 years old
* Indicated for elective periacetabular osteotomy

Exclusion Criteria:

* Preoperative use of an anticoagulant (Plavix, warfarin, lovenox, etc.)
* History of hypersensitivity to tranexamic acid
* History of thromboembolic event (e.g., Pulmonary embolism or Deep vein thrombosis)
* History of subarachnoid hemorrhage
* History or evidence of hepatic dysfunction (aspartate transaminase-alanine transaminase ratio greater than 60) or renal dysfunction (Creatinine greater than 1.5 mg/dL, or glomerular filtration rate less than 30 mL/minute)
* History of seizure
* Coronary stents or prior diagnosis of coronary artery disease
* Color blindness
* Leukemia
* Congenital or acquired coagulopathy as evidence by international normalized ratio (INR) greater than 1.4 or partial thromboplastin time (PTT) > 1.4 times normal, or Platelets less than 150,000/mm^3 on preoperative laboratory testing
* Use of hormone replacement therapy or hormonal contraceptive agent within 7 days prior to surgery
* Pregnant
* Breastfeeding
* Donated preoperative autologous blood
* Younger than 12-years-old and older than 45-years-old
* Preoperative hemoglobin less than 10 g/dL
* Concomitant open procedures (e.g., femoral osteotomy or osteochondral allograft)
* Patients with any contraindication to neuraxial anesthesia:
* Patient refusal
* History of lumbar spinal fusion
* Infection at the site of the epidural
* Coagulopathy, as defined above
* Ventriculoperitoneal shunt

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest L. Sink, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: Patients randomized to this arm will receive standard dosing of tranexamic acid intraoperatively.
  Tranexamic Acid
- Placebo: Patients randomized to this arm will receive normal saline solution, instead of tranexamic acid, intraoperatively.
  Placebo
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 45 | 44
Completed | 40 | 41
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Unknown concomitant procedure | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 16
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (7.2) | 26.8 (7.7) | 25.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Calculated Total Blood Loss
Description: Calculated total blood loss by patients
Time Frame: 1day (Hospital Admission)
Measure: Mean (Full Range); unit: mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 40 | 41
mL | 1264.6 [483.6 to 2046.9] | 1515.4 [724.7 to 2582.2]

2. Secondary Outcome: Number of Patients With Allogenic Blood Transfusion
Description: Total allogenic blood transfusion
Time Frame: 1day (Hospital Admission)
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 40 | 41
participants | 4 | 15

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, up to 6 weeks
Description: Only serious venous thromboembolic complications were monitored/assessed.
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02253810/Prot_SAP_000.pdf